CLINICAL TRIAL: NCT00967200
Title: Identification of Genes Involved in the Pathogenesis of Gliomas by Transcriptome Analysis
Brief Title: Study of Tissue Samples From Patients With Glioma or Other Brain Tumors
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 7745
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Central Nervous System Lymphoma
Keywords: adult anaplastic astrocytoma; adult diffuse astrocytoma; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma; adult pilocytic astrocytoma; adult pineal gland astrocytoma; adult subependymal giant cell astrocytoma; adult brain stem glioma; adult choroid plexus tumor; adult craniopharyngioma; adult ependymoblastoma; adult medulloblastoma; adult supratentorial primitive neuroectodermal tumor (PNET); adult anaplastic ependymoma; adult ependymoma; adult myxopapillary ependymoma; adult subependymoma; meningeal melanocytoma; adult meningeal hemangiopericytoma; adult grade I meningioma; adult grade II meningioma; adult anaplastic meningioma; adult papillary meningioma; adult anaplastic oligodendroglioma; adult oligodendroglioma; adult pineoblastoma; adult pineocytoma; adult mixed glioma; recurrent adult brain tumor
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Gliosarcoma; Choroid Plexus Neoplasms; Craniopharyngioma; Neuroectodermal Tumors, Primitive; Medulloblastoma; Ependymoma; Glioma, Subependymal; Meningioma; Oligodendroglioma; Pinealoma; Glioma; Brain Neoplasms | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: laboratory biomarker analysis — laboratory biomarker analysis
Other: pharmacogenomic studies — pharmacogenomic studies

SUMMARY:
RATIONALE: Studying the genes expressed in samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at tissue samples from patients with glioma or other brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To better understand the pathophysiology of gliomas and identify molecular markers that may predict prognosis and progression or that could identify new therapeutic approaches.

Secondary

* To compare gene expression profiles, in terms of response to treatment, and attempt to isolate subgroups of patients with objective response to certain types of chemotherapy or radiotherapy.

OUTLINE: This is a multicenter study.

Biological samples are collected from patients at time of surgery for diagnostic and/or treatment purposes.

ELIGIBILITY:
Inclusion Histologically confirmed glioma of any grade or rare primary brain tumor No urgent situation No known or suspected active infection Must not be deprived of liberty or protected by law Not pregnant or nursing

Exclusion :

No concurrent participation in other trials that require a period of exclusion

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathophysiology of gliomas and identification of molecular markers that may predict prognosis and progression or that could identify new therapeutic
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2003-11; Primary Completion 2009-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pathophysiology of gliomas | 1 day
  Pathophysiology of gliomas that may predict prognosis and progression or that could identify new therapeutic

SECONDARY OUTCOMES:
Identification of molecular | 1 day
  Identification of molecular markers that may predict prognosis and progression or that could identify new therapeutic

CONTACTS AND LOCATIONS:
Overall Officials: Luc Bauchet, MD, Principal Investigator — University Hospital, Montpellier
Locations (2):
- France (2):
  - CHU Montpellier, Montpellier
  - Clinique Gui de Chauliac, Montpellier